CLINICAL TRIAL: NCT00728845
Title: (NJ 1508) Modulation of Autophagy With Hydroxychloroquine in Combination With Carboplatin, Paclitaxel and Bevacizumab in Patients With Advanced/Recurrent Non-Small Cell Lung Cancer - A Phase I/II Study
Brief Title: Hydroxychloroquine, Carboplatin, Paclitaxel, and Bevacizumab in Recurrent Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000600241; P30CA072720 (NIH); CINJ-030801 (Other: CINJ); NCT00933803 (obsolete NCT alias)
Record Dates: First submitted 2008-08-05; First posted 2008-08-06 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; large cell lung cancer; recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Hydroxychloroquine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab (Experimental): Cohort 1: Bevacizumab Eligible Patients All on Day 1 Paclitaxel 200mg/m2 IV over 3 hours Carboplatin AUC= 6 IV over 15-30 min Bevacizumab 15 mg/kg IV over 90 min for PLUS Hydroxychloroquine 200 mg PO BID Cycles every 3 weeks for 4-6 Cycles
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: hydroxychloroquine; Drug: paclitaxel
- Hydroxychloroquine, Carboplatin, Paclitaxel (Experimental): Cohort 2: Bevacizumab Ineligible Patients All on Day 1 Paclitaxel 200mg/m2 IV over 3 hours Carboplatin AUC= 6 IV over 15-30 min PLUS Hydroxychloroquine 200 mg PO BID Cycles every 3 weeks for 4-6 Cycles
  Interventions: Drug: carboplatin; Drug: hydroxychloroquine; Drug: paclitaxel

INTERVENTIONS:
Biological: bevacizumab — Only patients eligible for bevacizumab will receive bevacizumab. Dose is at 15 mg/kg on day 1 of each cycle.
  Arms: Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab
Drug: carboplatin — Carboplatin will be given at AUC = 6 by IV over 15-30 minutes on Day 1 immediately following paclitaxel
Drug: hydroxychloroquine — 200 mg orally BID (total daily dose of 400 mg)
Drug: paclitaxel — Dose of 200 mg/m2 IV on day 1 of each cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as hydroxychloroquine, carboplatin, and paclitaxel and work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving hydroxychloroquine together with carboplatin, paclitaxel and bevacizumab may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of hydroxychloroquine when given together with carboplatin, paclitaxel, and bevacizumab and to see how well they work in treating patients with recurrent advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the recommended phase II dose of hydroxychloroquine and carboplatin in combination with paclitaxel and bevacizumab in patients with advanced recurrent non-small cell lung cancer. (Phase I)
* To assess the antitumor activity, as measured by tumor response rate, of this regimen in these patients. (Phase II)

Secondary

* To measure time to progression, progression-free survival, and overall survival of these patients.
* To assess the incidence of toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. This is a phase I, dose-escalation study of carboplatin and hydroxychloroquine followed by a phase II study.

Patients receive paclitaxel IV over 3 hours, carboplatin IV over 15-30 minutes, and bevacizumab IV over 90 minutes on day 1 and oral hydroxychloroquine on days 1-21. Treatment repeats every 21 days for a total of 4 courses. Patients then receive bevacizumab IV over 30-90 minutes every 21 days and oral hydroxychloroquine daily for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced non-small cell lung cancer, meeting the following criteria:

  * Recurrent disease
  * No component of squamous cell carcinoma
  * Mixed tumors will be categorized by predominant cell type

    * No mixed histology with small cell component
* Diagnosis established on metastatic tumor aspirate or biopsy (not sputum cytology alone) and meets 1 of the following staging criteria:

  * Stage IIIB disease with malignant pleural effusion
  * Stage IV disease
* Measurable disease
* More than 1 year since post-operative adjuvant therapy for previously resected non-small cell lung cancer with evidence of disease progression
* No known CNS metastases by CT scan or brain MRI within the past 28 days

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) (≤ 2 times ULN and no other liver function test abnormality in patients with Gilbert disease)
* AST/ALT ≤ 2.5 times ULN (≤ 5 times ULN in the presence of liver metastases)
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* INR ≤ 1.5 and aPTT normal
* Urine protein:creatinine ratio < 1.0 OR urine protein ratio < 1,000 mg by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection
* No psoriasis or porphyria
* No HIV positivity
* No significant traumatic injury within the past 28 days
* No serious non-healing wound, ulcer, or bone fracture
* No peripheral or sensory neuropathy > grade 1
* No hypertension that cannot be controlled by antihypertensive medication (i.e., blood pressure > 150/100 mm Hg despite optimal medical therapy)
* No cardiovascular disease, including any of the following:

  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * History of significant vascular disease (e.g., aortic aneurysm)
  * Symptomatic peripheral vascular disease within the past 6 months
  * Myocardial infarction within the past 6 months
  * Stroke within the past 6 months
* No other active malignancy within the past 3 years, except curatively treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or ductal or lobular carcinoma in situ of the breast, or other curatively treated malignancy with no evidence of disease > 3 years
* No retinal or visual field changes from prior 4-aminoquinoline compound therapy
* No known hypersensitivity to 4-aminoquinoline compound
* No known glucose-6-phosphate (G-6P) deficiency
* No known bleeding diathesis or coagulopathy
* No known gastrointestinal pathology that would interfere with drug bioavailability
* No known prior hypersensitivity to carboplatin, paclitaxel, bevacizumab, hydroxychloroquine, or any of their components
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No history of gross hemoptysis (i.e., bright red blood of a ½ teaspoon or more) within the past 3 months
* No history of any social or medical condition that, in the investigator's opinion, might interfere with the patient's ability to comply with the protocol or pose additional or unacceptable risk to the patient

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior radiation to sites other than the brain, and recovered to ≤ grade 1
* At least 28 days since prior and no concurrent full-dose anticoagulants or thrombolytic agents
* At least 28 days since prior major surgical procedure or open biopsy and no anticipated need for such during study therapy

  * Vascular access device placement with wound recovery allowed before study
* No prior cytotoxic chemotherapy or targeted therapy in the advanced or metastatic setting
* No concurrent treatment for rheumatoid arthritis or systemic lupus erythematosus
* No concurrent combination antiretroviral therapy
* No concurrent hydroxychloroquine for treatment or prophylaxis of malaria
* No concurrent aurothioglucose
* No other concurrent investigational or commercial agent or therapy for this malignancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-06-16 (Actual); Primary Completion 2010-12-21 (Actual); Study Completion 2010-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Aisner, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/show/NCT00728845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Cancer Institute of New Jersey (a comprehensive cancer center) and the Robert Wood Johnson University Hospital-Hamilton in New Jersey from June 2008 through December 2010.
Period: Overall Study
Arm/Group | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab | Hydroxychloroquine, Carboplatin, Paclitaxel
Started | 8 | 0
Completed | 8 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab | Hydroxychloroquine, Carboplatin, Paclitaxel | Total
Number analyzed (Participants) | 8 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 4 |  | 4
  >=65 years | 4 |  | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (8.4) |  | 63.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 5 |  | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose of Hydroxychloroquine and Carboplatin When Administered With Paclitaxel and Bevacizumab (Phase I)
Time Frame: Followed for the duration of the phase 1 treatment, an average of 18 weeks
Population: Study was terminated early and insufficient data were collected to assess this outcome measure.
Arm/Group | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab | Hydroxychloroquine, Carboplatin, Paclitaxel
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Overall Response (Phase II)
Time Frame: Treatment start date to date of best response
Population: Study was terminated early and insufficient data were collected to assess this outcome measure.
Arm/Group | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab | Hydroxychloroquine, Carboplatin, Paclitaxel
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Progression (Phase II)
Time Frame: Treatment start date and date of progression
Population: Study was terminated early and insufficient data were collected to assess this outcome measure.
Arm/Group | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab | Hydroxychloroquine, Carboplatin, Paclitaxel
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression-free Survival at 1 Year (Phase II)
Time Frame: Treatment start date to 1 year
Population: Study was terminated early and insufficient data were collected to assess this outcome measure.
Arm/Group | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab | Hydroxychloroquine, Carboplatin, Paclitaxel
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (Phase II)
Time Frame: Treatment start date to date of death
Population: Study was terminated early and insufficient data were collected to assess this outcome measure.
Arm/Group | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab | Hydroxychloroquine, Carboplatin, Paclitaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years and 6 months
Arm/Group | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab | Hydroxychloroquine, Carboplatin, Paclitaxel
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab (N=8) | Hydroxychloroquine, Carboplatin, Paclitaxel (N=0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine, Carboplatin, Paclitaxel, Bevacizumab (N=8) | Hydroxychloroquine, Carboplatin, Paclitaxel (N=0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 7 (13) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6 (15) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 5 (9) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 4 (8) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Anorexia (Gastrointestinal disorders) | 3 (4) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 0 (0)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 7 (16) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 0 (0)
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Mood alteration - Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Neuropathy: motor (Psychiatric disorders) | 1 (1) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 5 (7) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain - Extremity-limb (General disorders) | 3 (5) | 0 (0)
Pain - Abdomen NOS (General disorders) | 2 (2) | 0 (0)
Pain - Bone (General disorders) | 2 (2) | 0 (0)
Pain - Chest wall (General disorders) | 2 (2) | 0 (0)
Pain - Chest/thorax NOS (General disorders) | 2 (2) | 0 (0)
Pain - Back (General disorders) | 1 (1) | 0 (0)
Pain - Buttock (General disorders) | 1 (1) | 0 (0)
Pain - Dental/teeth/peridontal (General disorders) | 1 (1) | 0 (0)
Pain - Head/headache (General disorders) | 1 (1) | 0 (0)
Pain - Joint (General disorders) | 1 (1) | 0 (0)
Pain - Oral cavity (General disorders) | 1 (1) | 0 (0)
Pain - Other (Specify, __) (General disorders) | 1 (1) | 0 (0)
Pain - Stomach (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (8) | 0 (0)
Weight loss (General disorders) | 5 (7) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (3) | 0 (0)
Insomnia (General disorders) | 2 (2) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 3 (3) | 0 (0)
Glucose, serum-high (hyperglycemia) (Investigations) | 3 (4) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 (2) | 0 (0)
Alkaline phosphatase (Investigations) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Investigations) | 1 (1) | 0 (0)
Metabolic/Laboratory - Other (Specify, __) (Investigations) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Investigations) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 5 (10) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3 (4) | 0 (0)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (General disorders) | 1 (1) | 0 (0)
Hemorrhage, GI - Upper GI NOS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage, GU - Bladder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection - Other (Specify, __) (Infections and infestations) | 2 (2) | 0 (0)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 1 (1) | 0 (0)
Edema: limb (Vascular disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes